CLINICAL TRIAL: NCT06977971
Title: Evaluation of Clinical, Laboratory, and Radiologic Parameters Affecting Antibiotic Use and Associated Cost in RSV-Positive Children With Acute Lower Respiratory Tract Infections
Brief Title: RSV Antibiotic Drivers And Resource-use
Acronym: RADAR
Status: Completed | Type: Observational
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Burcu Busra Acar, Pediatric Cardiology Fellow, Ege University Faculty of Medicine, Dr. Behcet Uz Children's Hospital
Other Study IDs: 2021-634
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Virus Infections; Antibiotic Stewardship in Community Hospitals
Keywords: Respiratory Syncytial Virus Infections; Anti-Bacterial Agents; Health Care Costs; Polymerase Chain Reaction; C-Reactive Protein
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RSV-Positive Children Aged 1-24 Months: This cohort includes children aged 1 to 24 months who were hospitalized with laboratory-confirmed RSV-positive acute lower respiratory tract infections between April 2017 and April 2021. Data were collected retrospectively at Dr. Behçet Uz Children's Hospital. No intervention was administered as part of the study; the investigation focused on clinical, laboratory, and radiologic factors influencing antibiotic use, as well as associated hospitalization costs.

SUMMARY:
This study retrospectively evaluated the clinical, laboratory, and radiologic factors that influence the decision to prescribe antibiotics in children under 2 years of age hospitalized with RSV-positive acute lower respiratory tract infections. The study also examined the economic impact of antibiotic use in these patients. The goal is to improve clinical decision-making and reduce unnecessary antibiotic exposure in children with viral infections.

DETAILED DESCRIPTION:
This retrospective, single-center study aimed to assess the clinical decision-making process regarding antibiotic prescription in children aged 1 to 24 months hospitalized with RSV-positive acute lower respiratory tract infections (ALRTI). The study was conducted at Dr. Behçet Uz Children's Hospital and covered four consecutive RSV seasons (April 2017 - April 2021). RSV infection was confirmed via multiplex PCR.

Clinical and laboratory variables potentially influencing antibiotic use included fever, respiratory distress, CRP levels, leukocyte count, and radiologic findings such as infiltrates on chest X-ray. The study also examined whether antibiotic selection (agent, timing, and duration) was associated with specific clinical profiles or severity indicators.

Hospitalization cost data were analyzed to estimate the economic burden of antibiotic use in RSV-positive patients. The study contributes to improved antimicrobial stewardship by identifying patterns of potentially unnecessary antibiotic prescriptions in viral respiratory infections.

Ethical approval was obtained from the local ethics committee (Approval No: 2021-634), and the study adhered to the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 24 months at the time of hospitalization
* Laboratory-confirmed RSV positivity via multiplex PCR
* Hospitalized for acute lower respiratory tract infection
* Complete hospitalization and clinical data available

Exclusion Criteria:

* Detection of additional respiratory pathogens on multiplex PCR
* Discharge against medical advice before treatment was completed
* Missing or incomplete key clinical, laboratory, or radiologic data
* ICU admission without full follow-up data

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalized children aged 1 to 24 months with laboratory-confirmed RSV-positive acute lower respiratory tract infections, treated at Dr. Behçet Uz Children's Hospital between April 2017 and April 2021.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Association between clinical/laboratory/radiologic parameters and antibiotic prescription | During hospitalization (April 2017 - April 2021)
  This outcome assesses the relationship between objective findings (e.g., CRP levels, abnormal chest X-ray, fever) and the decision to initiate antibiotic therapy in RSV-positive children aged 1-24 months hospitalized with acute lower respiratory tract infections.

SECONDARY OUTCOMES:
Total antibiotic-related hospitalization cost per patient | During hospitalization (April 2017 - April 2021)
  This outcome evaluates the economic impact of antibiotic use by calculating the direct hospitalization costs associated with antibiotic treatment in RSV-positive pediatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Büşra B Acar, Pediatric Cardiology Fellow, Principal Investigator — Ege University; Burcu Büşra B Acar, Pediatric Cardiology Fellow, Principal Investigator — Ege University Faculty of Medicine, Department of Pediatric Cardiology
Locations (1):
- Dr. Behçet Uz Children's Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study is a retrospective observational analysis based on de-identified hospital records. Individual participant data will not be shared due to ethical considerations and the absence of participant consent for data sharing.

DOCUMENTS (2):
  • Study Protocol (2025-05-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT06977971/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT06977971/SAP_001.pdf